CLINICAL TRIAL: NCT06622629
Title: NATURE-based Therapy in Urban Coast in Barcelona (NATURE-MET-B)
Brief Title: Nature Based Therapy With Mindful Walks in Urban Coastal Setting - Barcelona (Spain)
Acronym: NATURE-MET-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/11524/I; 101081420 RESONATE (Other Grant/Funding Number: HORIZON-CL6-2022-COMMUNITIES-02-two-stage)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: social prescription; Social-ecological system; stress; quality of life; blue health; resilience; nature based therapy
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Grop (Experimental): * Adults aged >=18 years
  * Smartphone users
  * Understand Spanish and/or Catalan language
  Interventions: Other: Nature based Therapy (NbT): Planned therapeutic techniques performed in natural settings and based on nature-human active participation and connection
- Control group (Active Comparator): * Adults aged >=18 years
  * Smartphone users
  * Understand Spanish and/or Catalan language The control group participants are assessed at the same time as those in the intervention group (t1, t2, and t3). Participants in the control group will be offered the opportunity to benefit from the NbT once the follow-up period is completed (day 70).
  Interventions: Other: Waiting List

INTERVENTIONS:
Other: Nature based Therapy (NbT): Planned therapeutic techniques performed in natural settings and based on nature-human active participation and connection — The intervention consists of a 5-week (35-day) conscious immersion treatment in a natural coastal urban environment, involving approximately three sessions per week of semi-structured walking and mindfulness exercises lasting 60 minutes. Following this, there will be a follow-up period that will end 5 weeks after the intervention has concluded (day 70). Participants will document and evaluate the therapy sessions at the location where the mindfulness exercises take place, using the mobile phone application App, a digital tool for assessing the environment and health. The aim is to integrate nature-based physical activity and relaxation sessions into daily life.
  The intervention will be standardized as much as possible to allow comparison of the results with those from the other study centers in Salzburg (Vienna) and Padua (Italy).
  Arms: Intervention Grop
Other: Waiting List — Participants in the control group will be offered the opportunity to benefit from the NbT once the follow-up period is completed (day 70).
  Arms: Control group

SUMMARY:
The main objective of the NATURE-MET-B (Barcelona) study is to analyze the effects of a Nature-based Therapy (NbT) on the biopsychological resilience of adults general population through changes in: i) health-related quality of life and ii) allostatic load (physiological stress). The secondary objective is to provide data on the environmental, social, and economic aspects of the intervention in order to refine specific prevention programs and establish programs that include NbT as a secondary preventive measure in healthcare.

Analogous to NATURE-MET-B, two similar NbT studies will be carried out in Padua (Italy) and Salzburg (Austria) for the secondary prevention of Metabolic Syndrom (MetS). These are not multicenter studies but three comparable studies with similar inclusion and exclusion criteria in all study locations. Only the types of landscape and natural exposure sites differ: Barcelona-Coastal Urban, Padua-Urban Green, Salzburg-Mountainous Rural.

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18 years
* Smartphone users

Exclusion Criteria:

* Acute contraindications

  - Malignant hypertension
* Contraindications or differential diagnosis

  * Severe respiratory or pulmonary disease (COPD, severe asthma, emphysema)
  * Arteriosclerotic incident (e.g., myocardial infarction) 6 months previous the study starting
  * Heart failure
  * Uncontrolled metabolic diseases (e.g., diabetes mellitus)
  * Diagnosis or treatment of a malignant disease < 3 years ago
  * Chronic immunological diseases (e.g., rheumatoid arthritis)
  * Orthopedic conditions that prevent participation in excursions
* Factors that prevent or hinder participation in the intervention program

  * Alcohol or substance abuse (except nicotine)
  * Pregnancy
  * Insufficient knowledge of Spanish or Catalan (written and spoken/questionnaires)
  * Factors that prevent self-management
  * Moderate to severe depression (score < 13 points on the WHO-5)
  * Other untreated severe psychiatric illnesses (e.g., schizophrenia)
  * Taking certain medications
  * Use of weight loss supplements
  * Participation in another clinical intervention trial
  * Participation in therapeutic weight loss programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (SF-12) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The SF-12 (Short Form 12) is a widely used survey instrument that measures health-related quality of life (HRQoL). It is a shorter version of the SF-36, designed to assess a person´s physical and mental health status through 12 questions. The SF-12 provides a quick and reliable means to evaluate the impact of health on an individual's quality of life, making it useful in clinical settings and research.
Allostatic Index-ALI | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Allostatic Index (ALI) is a biomarker-based measure designed to assess the cumulative physiological burden of stress on the body over time. It reflects the wear and tear on the body caused by chronic stress and the body's response to it, offering insights into an individual's health status and risk for various diseases.
Scale of Positive and Negative Experience (SPANE) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Scale of Positive and Negative Experience (SPANE) is a brief, self-report measure designed to assess an individual's emotional experiences over a specified period. SPANE provides insights into both positive and negative feelings, contributing to the broader understanding of subjective well-being and emotional health.

SECONDARY OUTCOMES:
Environmental Concerns | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  Environmental Concerns (adapted from W. Schultz, 2001) refers to a psychological framework designed to measure the extent and type of concerns individuals have regarding environmental issues. The original framework by Wesley Schultz distinguishes between different types of environmental concerns based on their underlying motivations and the values driving them.
  The adapted Environmental Concerns Scale often uses a Likert scale (e.g., from 1 = "not concerned at all" to 5 = "extremely concerned") to assess how strongly individuals resonate with each type of concern. This helps identify whether a person is more motivated by personal impacts, the well-being of others, or the intrinsic value of nature.
Revised Pro-Environmental Behavior Scale (R-PEBS) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Revised Pro-Environmental Behavior Scale (R-PEBS) is a psychometric tool used to measure the frequency and extent of individuals' engagement in behaviors that promote environmental sustainability. The scale helps identify specific actions that people take in their daily lives to reduce their ecological footprint and contribute to environmental conservation. The revised version aims to improve clarity and relevance, adapting to modern environmental challenges.
  Respondents typically rate their frequency of engaging in these behaviors using a Likert scale (e.g., from 1 = "never" to 5 = "always"). The total score reflects the individual's overall level of pro-environmental behavior. Higher scores suggest a greater commitment to sustainability and ecological responsibility.
Quality-Adjusted Life Years (QUALYs) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  (QUALYs) is a measure used to evaluate the value of health outcomes by considering both the quantity (years of life) and quality of life. It's a widely used metric in health economics, especially for cost-effectiveness analyses of healthcare interventions. QUALYs combine life expectancy with a weighting factor representing the quality of life during those years, where 1 represents perfect health and 0 represents death.
Healthcare and Social System Utilization (Cost Savings) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  Healthcare and social system utilization refers to the frequency and types of services used by individuals, while cost savings in this context involves reducing the financial burden on these systems through efficient resource use, preventive measures, or improved treatment outcomes. Cost savings in healthcare and social services can be measured through reduced hospital visits, fewer medications, shorter hospital stays, or less reliance on long-term care services.
  The primary aim of assessing healthcare utilization and cost savings is to analyze how specific interventions or programs (such as lifestyle changes, treatments, or preventive health measures) can improve health outcomes while reducing the costs incurred by the healthcare and social systems.
Willingness to Pay (WTP) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  Willingness to Pay (WTP) refers to the maximum amount an individual is willing to pay for a specific good or service, reflecting their perceived value of that item. In health economics, WTP is often used to gauge how many individuals value health improvements, treatments, or healthcare interventions.
Nature Connectedness Index (NCI) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Nature Connectedness Index (NCI) is a psychological measure designed to assess an individual's emotional and cognitive relationship with nature. This index is rooted in the idea that a strong connection to nature is beneficial for mental health, well-being, and environmental behavior. By measuring nature connectedness, researchers and practitioners can better understand the impact of nature on individual and community health.
Five Facet Mindfulness Questionnaire- FFMQ-15 | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Five Facet Mindfulness Questionnaire (FFMQ) is a widely used self-report instrument designed to assess mindfulness-a mental state characterized by focused attention, awareness, and acceptance of the present moment. The FFMQ-15 is a shorter version of the original FFMQ, which consists of 39 items. The 15-item version provides a concise yet effective means of evaluating mindfulness across five key dimensions
State-Trait-Assessment of Resilience Scale (STARS) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The State-Trait Assessment of Resilience Scale (STARS) is a psychological tool designed to measure resilience in individuals. Resilience refers to the capacity to adapt and thrive in the face of adversity, stress, or trauma. The STARS framework differentiates between two aspects of resilience: state resilience, which reflects an individual's current ability to cope with stress, and trait resilience, which indicates a more stable, enduring characteristic of resilience over time
Perceived Stress Scale (PSS) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Perceived Stress Scale (PSS) is a widely used psychological instrument designed to measure the perception of stress in individuals. The PSS assesses how unpredictable, uncontrollable, and overloaded individuals perceive their lives to be. It helps researchers and clinicians understand how stress impacts mental and physical health.
  The PSS consists of a series of questions that assess various aspects of perceived stress over a specific time frame (usually the past month). The PSS can be administered in different versions, commonly consisting of 10 or 14 items. Participants respond using a 5-point Likert scale (0-4). Th scores for each item are summed to produce a total score, which can range from 0 to 40 (in the 10-item version) or up to 56 (in the 14-item version). Scores can be categorized into ranges (e.g., low, moderate, high stress) to help assess individuals' stress. Higher scores indicate higher levels of perceived stress.
Subjective well-being and quality of life-OCDE-4 | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The OECD-4 refers to a set of four indicators used by the Organisation for Economic Co-operation and Development (OECD) to assess subjective well-being and quality of life among individuals and populations. This framework aims to provide a comprehensive understanding of well-being beyond traditional economic measures, focusing instead on people's perceptions of their lives.
  The OECD-4 indicators provide a valuable framework for assessing subjective well-being and quality of life. By focusing on life satisfaction, positive and negative feelings, and overall health, the OECD-4 offers insights into individuals' perceptions of their lives and well-being.
De Jong Gierveld Loneliness Scale | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The De Jong Gierveld Loneliness Scale is a psychological tool designed to assess feelings of loneliness in individuals. Developed by Dutch psychologist Jenny de Jong Gierveld in the 1980s, this scale distinguishes between emotional and social loneliness, making it a comprehensive measure of loneliness in various contexts.
Brief Sense of Community Scale (BSCS) | From starting to the end of the intervention (5 weeks)
  The Brief Sense of Community Scale (BSCS) is a psychological instrument designed to measure individuals' feelings of belonging and connection within a community. Developed by Chavis, Hogge, McMillan, and Wandersman in the 1980s, the scale has been widely used in various research contexts to assess the sense of community in different populations.The BSCS typically uses a Likert-type scale for responses. Components of the Brief Sense of Community Scale: Belonging, membership, emotional connection, common values.
Social Desirability Scale - Short Form | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Social Desirability Scale - Short Form is a condensed version of scales designed to measure social desirability bias, which is the tendency of respondents to answer questions in a manner that will be viewed favorably by others. This short form allows for efficient assessment of social desirability without requiring extensive time or effort from participants.
  Components: Positive Self-Presentation, Avoidance of Negative Trait.The Short Form often uses a Likert-type scale for responses (1-5)
Self-Determined Motivation Scale (SDMS) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Self-Determined Motivation Scale (SDMS) is an assessment tool used to measure the levels and types of motivation in individuals, particularly within educational, occupational, and sports contexts. This scale is based on Self-Determination Theory (SDT), which differentiates between various forms of motivation, from intrinsic to extrinsic, and emphasizes the importance of autonomy and self-regulation in fostering optimal motivation and well-being.
  Components:Intrinsic Motivation, Extrinsic Motivation, Motivation. The SDMS typically employs a Liker-type scale for responses, often using a range from 1 to 7
Ideal Self | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Ideal Self is a psychological construct that represents the person one aspires to become. It encompasses traits, values, and achievements that individuals perceive as desirable and motivating. According to Ganesan (2020), understanding and aligning one's behaviors with the ideal self can lead to greater satisfaction and motivation in various aspects of life.
  Components:Personal Values, Goals and Aspirations, Self-Perception, Emotional and Psychological Well-Being, Behavioral Alignment
Perception of local nature (PANS-6) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Perception of Local Nature Scale (PANS-6) is a measurement tool designed to assess individuals' perceptions and feelings about the natural environment in their local area. This scale focuses on how people view and relate to the nature around them, which can impact their well-being, environmental behaviors, and sense of connection to the natural world. The PANS-6 typically consists of six items that capture various dimensions of the perception of local nature. These items may focus on aspects such as: Appreciation, Sense of Connection, Quality of Experience, Accessibility, Biodiversity Awareness, motional Response.The PANS-6 often employs a Likert-type scale for responses, where participants indicate their level of agreement with each statement (1-5)
Environmental Attitudes/Environmental concerns | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Environmental Concerns Scale is a measurement tool that assesses individuals' concerns regarding environmental issues. Adapted from the work of W. Schultz (2001), this scale focuses on various dimensions of environmental awareness and attitudes, exploring how these concerns influence behaviors and attitudes toward environmental protection and sustainability.The scale typically consists of several items that cover various aspects of environmental concerns, which may include: Global Environmental Issues, Local Environmental Issues, Personal Impact, Responsibility and Action, Future Generations.The Environmental Concerns Scale usually employs a Likert-type scale for responses, where participants indicate their level of agreement or concern regarding each statement (1-5)
Perceived Restorativeness Scale (PRS) | From starting to the end of the intervention (5 weeks)
  The Perceived Restorativeness Scale (PRS) is a psychological tool designed to assess the restorative qualities of environments, particularly natural and green spaces. Developed by Hartig, Korpela, and Staats (2003), the PRS evaluates how certain environments facilitate recovery from mental fatigue and stress, contributing to overall well-being and restoration.The PRS typically consists of several items that capture key dimensions of perceived restorativeness, including: Fascination, Being Away, Extent,Compatibility. The PRS often uses a Likert-type scale for responses, where participants indicate their level of agreement with each statement (1-5)
Five Facet Mindfulness Questionnaire- FFMQ-15 | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The Five Facet Mindfulness Questionnaire (FFMQ-15) is a shortened version of the original FFMQ designed to assess various aspects of mindfulness. Developed by Baer et al. (2006), this questionnaire evaluates how individuals relate to their thoughts and feelings in a way that allows for greater awareness and acceptance. It is widely used in both research and clinical settings to explore the impact of mindfulness on mental health and well-being.The FFMQ-15 comprises 15 items that assess five facets of mindfulness: Observing, Describing, Acting with Awareness, Nonjudging of Inner Experience, Nonreactivity to Inner Experience.The FFMQ-15 uses a Likert-type scale for responses, where participants rate how true each statement is for them (1-5)
International Physical Activity Questionnaire (IPAQ - Short Form) | From enrollment to the end of treatment of treatment (5 weeks) and follow up (10 weeks)
  The International Physical Activity Questionnaire (IPAQ - Short Form) is a widely used tool for measuring physical activity levels in adults. Developed by a collaborative effort involving researchers from various countries, the IPAQ aims to provide a standardized method to assess the physical activity behaviors of individuals across different cultures and settings.The IPAQ - Short Form consists of several questions designed to capture different aspects of physical activity, including:Walking, Moderate-Intensity Physical Activity, Vigorous-Intensity Physical Activity, Sitting Time.The responses typically include options for frequency (days per week) and duration (minutes per day) for each type of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- ISGlobal, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Adequate measures will be implemented to ensure the protection and confidentiality of personal data, in accordance with Regulation (EU) 2016/679 on the Protection of Individuals with Regard to the Processing of Personal Data and on the Free Movement of Such Data, and Organic Law 3/2018, of December 5, on Personal Data Protection and the Guarantee of Digital Rights. National regulations on personal data protection will be implemented to ensure the highest standards in personal data management.
  Legality, fairness, and transparency; purpose limitation of processing; data minimization (only the necessary and relevant data for the research purpose will be collected); accuracy; storage limitation; and integrity and confidentiality will be applied when processing personal data. Personal data will not be transferred, except in cases permitted by law. Results will refer to analyses of aggregated data, no individual names will be associated with any published or unpublished report.
Supporting Information: Study Protocol